CLINICAL TRIAL: NCT01818323
Title: Phase I Trial: T4 Immunotherapy of Head and Neck Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, John Maher, Consultant and Senior Lecturer in Immunology, King's College London
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-001654-25
Record Dates: First submitted 2013-03-19; First posted 2013-03-26 (Estimated); Last update posted 2024-10-09 (Actual); Status verified 2024-03

CONDITIONS: Head and Neck Cancer
Keywords: Chimeric antigen receptor; Immunotherapy; Head and Neck Cancer; Phase I trial; Maximum tolerated dose
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: In this dose escalation study, the intervention consists of intratumoral delivery of panErbB-specific CAR T cells, administered alone or following lymphodepleting chemotherapy with fludarabine and cyclophosphamide. In cohort 7, patients will also receive 3 doses of Nivolumab, the first of which is administered 24h before CAR T-cells
  This note has been added in response to the warning " WARNING: Phase 1/Phase 2 studies typically have at least one Intervention Type of Drug, Biological/Vaccine or Combination Product."
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intra-tumoral T4 immunotherapy (Experimental): Treatment arms comprise escalating doses of T4 immunotherapy, administered alone or in combination with lymph-depleting chemotherapy
  Interventions: Other: Intra-tumoral T4 immunotherapy

INTERVENTIONS:
Other: Intra-tumoral T4 immunotherapy — Intra-tumoral administration of a single dose of T4-positive patient-derived T-cells (at five escalating dose levels) contained within 1-4 mL. Cohort 6 patients receive CAR T-cells (dose level 3) after lymphodepletion with fludarabine and cyclophosphamide. Cohort 7-8 patients receive T4 cells after lymphodepletion as above, combined with 4 doses of nivolumab.
  Other Names: 4ab T1E28z positive T-cells

SUMMARY:
The overall goal of this study is to investigate the safety of T4 immunotherapy when administered to treat loco-regional disease in Squamous Cell Cancer of the Head and Neck (SCCHN) that is not suitable for conventional active therapy.

The investigators propose to conduct an open-labelled, non-randomized, dose-escalation phase I trial in which autologous T4+ T-cells are administered to patients with SCCHN. T-cells will be engineered to express a second generation chimeric antigen receptor (CAR) named T1E28z. Engineered T-cells will be injected directly into the tumour site. Patients will not be lymphodepleted. A classical 3+3 design will be employed, with dose escalation from 10^7 through to 10^9 transduced T4+ T-cells, dependent upon toxicity monitoring. It is anticipated that up to 30 patients will be enrolled over the course of the study.

DETAILED DESCRIPTION:
Further information is provided in van Schalkwyk MC, Papa SE, Jeannon JP, Guerrero Urbano T, Spicer JF, Maher J. Design of a phase I clinical trial to evaluate intratumoral delivery of ErbB-targeted chimeric antigen receptor T-cells in locally advanced or recurrent head and neck cancer. Hum Gene Ther Clin Dev. 2013 Sep;24(3):134-42. doi: 10.1089/humc.2013.144. PubMed ID: 24099518

ELIGIBILITY:
Inclusion Criteria:

1. Histologically and/ or cytologically confirmed SCCHN.
2. 18 years or older.
3. Locally advanced and/ or recurrent head and neck cancer with or without metastatic disease (excluding brain metastases) for whom no standard therapy remains or is suitable.
4. Regarding previous treatment, patients may have received prior systemic therapy, including platinum chemotherapy, at least one month earlier. In the presence of metastatic disease, recent short-course palliative radiotherapy to non-target site(s) is allowed.
5. Those who refuse palliative treatment may be eligible for participation. However, their reasons for not opting for palliative treatment must be explored thoroughly.
6. At least one loco-regional target lesion measurable by RECIST v1.1 criteria on CT or MRI scanning within four weeks of enrolment, and amenable to intra-tumoral injection.
7. Eastern Co-operative Oncology Performance Status of 0-2.
8. Normal cardiac function as assessed by electrocardiography and either echocardiography (ECHO), or multi-gated acquisition (MUGA) scanning. Left ventricular ejection fraction must be > 50%. Assessment must take place within four weeks of enrolment.
9. Haematology results within seven days of enrolment: neutrophils >1.5 x 109/L, platelets >100 x 109/L, haemoglobin >9g/dl, INR <1.5.
10. Biochemistry results within seven days of enrolment: • serum creatinine <1.5 upper limit of normal • bilirubin <1.25 times normal; • ALT/ AST <2.5 times upper limit of normal (<5 times upper limit of normal if liver metastases present)
11. Female patients must be postmenopausal (12 months of amenorrhea), surgically sterile or they must agree to use a physical method of contraception. Oral or injectable contraceptive agents cannot be the sole method of contraception. Women of childbearing potential (WOCB) who receive cyclophosphamide must adhere to these contraceptive requirements during the trial and until 3 months after the last dose of cyclophosphamide. Male patients, even if sterilized, must agree to use a barrier method of contraception. Male subjects must also commit to use a barrier method of contraception until at least 3 months after the end of study treatment.
12. Written informed consent prior to registration.
13. Eligible for NHS care in the UK.

Exclusion Criteria:

1. The presence of or imminent occurrence of airway obstruction, unless tracheostomy in place.
2. The presence of or imminent occurrence of tumour-mediated infiltration of major blood vessels.
3. Positive history of HIV-1, HIV-2, HTLV-1, HTLV-2, Hepatitis B, Hepatitis C or syphilis infection.
4. Prior splenectomy.
5. Clinically active autoimmune disease. Sub-clinical or quiescent autoimmune disease does not exclude from participation.
6. Treatment in the preceding week with systemic corticosteroids (> 20mg prednisolone/ day), any systemic immunomodulatory agent, radiotherapy, chemotherapy or investigational medicinal product.
7. Concurrent use of anticoagulant therapy is not permissible.
8. The presence of major co-morbidity likely to impair ability to undergo trial therapy, such as recent myocardial infarction, congestive cardiac failure or uncontrolled hypertension.
9. The presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
10. Cyclophosphamide allergy (Cohort 6 only).
11. Pregnancy.
12. Breastfeeding.
13. Prior T4 immunotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-06; Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities for T4 immunotherapy in SCCHN and determine a safe and feasible recommended dose for phase II testing of intra-tumoral T4 immunotherapy. | Up to 6 weeks post T4 administration
  Patients will be monitored intensely for the first 24 hours post T4 administration. Patients will the be assessed for signs of toxicity on days 3-4, 5-7, 8, 15, 29 and 43.

SECONDARY OUTCOMES:
To investigate serum cytokine levels after administration of T4 immunotherapy | up to 6 weeks post T4 administration
To investigate persistence of T4+ T-cells at the site of administration and in the peripheral circulation | up to 6 weeks post T4 administration
To achieve preliminary assessment of anti-tumour activity, using cross-sectional imaging to quantify objective responses | up to 6 weeks post T4 administration
To investigate tumour ErbB receptor phenotype, before and after administration of T4 immunotherapy | up to 6 weeks post T4 administration
To investigate immunomodulatory effects of metronomic cyclophosphamide on T4 immunotherapy | up to 6 weeks post T4 administration
  Pre- and post-treatment absolute number of circulating T-regulatory cells will be compared.
To investigate effect of T4 immunotherapy upon immune reactivity against endogenous tumour antigens | up to 6 weeks post T4 administration
  ELISPOT will be performed on blood samples taken 3 days prior and 29 days after T4 administration to measure for MAGE-reactive T-cells.

CONTACTS AND LOCATIONS:
Overall Officials: John Maher, MD PhD, Principal Investigator — King's College London
Locations (1):
- Clinical Research Facility, Guy's Hospital, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Davies DM, Foster J, Van Der Stegen SJ, Parente-Pereira AC, Chiapero-Stanke L, Delinassios GJ, Burbridge SE, Kao V, Liu Z, Bosshard-Carter L, Van Schalkwyk MC, Box C, Eccles SA, Mather SJ, Wilkie S, Maher J. Flexible targeting of ErbB dimers that drive tumorigenesis by using genetically engineered T cells. Mol Med. 2012 May 9;18(1):565-76. doi: 10.2119/molmed.2011.00493. PMID 22354215
- [Background] Wilkie S, Burbridge SE, Chiapero-Stanke L, Pereira AC, Cleary S, van der Stegen SJ, Spicer JF, Davies DM, Maher J. Selective expansion of chimeric antigen receptor-targeted T-cells with potent effector function using interleukin-4. J Biol Chem. 2010 Aug 13;285(33):25538-44. doi: 10.1074/jbc.M110.127951. Epub 2010 Jun 18. PMID 20562098
- [Background] van Schalkwyk MC, Papa SE, Jeannon JP, Guerrero Urbano T, Spicer JF, Maher J. Design of a phase I clinical trial to evaluate intratumoral delivery of ErbB-targeted chimeric antigen receptor T-cells in locally advanced or recurrent head and neck cancer. Hum Gene Ther Clin Dev. 2013 Sep;24(3):134-42. doi: 10.1089/humc.2013.144. PMID 24099518